CLINICAL TRIAL: NCT01345149
Title: Effect of Lifestyleintervention With Diet and Physical Activity in Obese Pregnant Women
Brief Title: Effect of Intervention With Diet and Physical Activity in Obese Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kristina Renault, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-D-2008-119
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Obesity
Keywords: Obesity; Pregnancy; Intervention; Diet; Physical activity
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diet + Exercise (Experimental): Diet: Intensive counselling about calorie restriction to reduce weight gain by dietician.
  Exercise: Individual counselling
  Interventions: Behavioral: Diet + Exercise
- Exercise (Experimental): Exercise: Individual counselling
  Interventions: Behavioral: Diet + Exercise
- Control (No Intervention): Standard treatment without intervention.

INTERVENTIONS:
Behavioral: Diet + Exercise — Diet: Intensive counselling about calorie restriction to reduce weight gain by dietician.
  Exercise: Individual counselling
  Other Names: Lifestyle intervention.
  Arms: Diet + Exercise; Exercise

SUMMARY:
Purpose: To evaluate if lifestyle intervention (diet and exercise) can reduce maternal weight gain, the incidence of pregnancy complications and minimize the number of macrosomic infants.

DETAILED DESCRIPTION:
Obese pregnant women with a BMI>30 are randomized to Diet + Exercise, Exercise or control (1:1:1) in order to reduce maternal weight gain to less than 5 kg during pregnancy.

The effect on the children of mothers in this study is evaluated in the study: Is it possible to reduce the Number of Macrosomic Infants With Abundant Fat Tissue by Lifestyle Intervention during Pregnancy (NCT01235676)

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* BMI > 30
* Singleton pregnancy
* Must speak and understand Danish

Exclusion Criteria:

* Alcohol or drug abuse
* Diabetes type I or other critical medical disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Maternal weight gain | At delivery, avarage 27 weeks after inclusion. For the last participant this will be aproximately April 2012

SECONDARY OUTCOMES:
Pregnancy complications | At delivery, avarage 27 weeks after inclusion. For the last participant this will be aproximately April 2012
Glucose tolerance in pregnancy | At delivery, avarage 27 weeks after inclusion. For the last participant this will be aproximately April 2012
Birth weight | At delivery, avarage 27 weeks after inclusion. For the last participant this will be aproximately April 2012

CONTACTS AND LOCATIONS:
Overall Officials: Niels Jørgen Secher, Professor, Study Chair — Department of Obstetrics and Gynecology, Hvidovre University Hospital; Lisbeth Nilas, Prof. DMSc, Study Chair — Department of Obstetrics and Gynecology, Hvidovre University Hospital
Locations (1):
- Department of Obstetrics and Gynecology, Hvidovre University Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Renault KM, Carlsen EM, Norgaard K, Nilas L, Pryds O, Secher NJ, Cortes D, Jensen JE, Olsen SF, Halldorsson TI. Intake of carbohydrates during pregnancy in obese women is associated with fat mass in the newborn offspring. Am J Clin Nutr. 2015 Dec;102(6):1475-81. doi: 10.3945/ajcn.115.110551. Epub 2015 Nov 11. PMID 26561621
- [Derived] Renault KM, Carlsen EM, Norgaard K, Nilas L, Pryds O, Secher NJ, Olsen SF, Halldorsson TI. Intake of Sweets, Snacks and Soft Drinks Predicts Weight Gain in Obese Pregnant Women: Detailed Analysis of the Results of a Randomised Controlled Trial. PLoS One. 2015 Jul 20;10(7):e0133041. doi: 10.1371/journal.pone.0133041. eCollection 2015. PMID 26192183